CLINICAL TRIAL: NCT02942303
Title: The Impact of Botulinum Toxin on Brow Height and Morphology: A Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, samer jabbour, MD, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USJ-03
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Brow Lifting
Keywords: Botulinum Toxin, Rejuvenation, Brow lift, Eyebrow.
MeSH Terms: interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Technique 1: Lateral orbicularis injections (Active Comparator): 5 equally spaced injections will be placed intramuscularly into the orbicularis under the lateral eyebrow starting lateral to the level of the lateral limbus and extending to the level of the inferior orbital rim.
  Interventions: Drug: Dysport; Procedure: lateral orbicularis injection
- 2. Technique 2: Lateral orbicularis and Corrugator injections (Active Comparator): 5 equally spaced injections will be placed intramuscularly into the orbicularis under the lateral eyebrow starting lateral to the level of the lateral limbus and extending to the level of the inferior orbital rim. In addition, 2 injections will be placed into the corrugator at the medial brow
  Interventions: Drug: Dysport; Procedure: Lateral orbicularis + corrugator injection

INTERVENTIONS:
Drug: Dysport
  Other Names: abobotulinumtoxineA
Procedure: lateral orbicularis injection
  Arms: Technique 1: Lateral orbicularis injections
Procedure: Lateral orbicularis + corrugator injection
  Arms: 2. Technique 2: Lateral orbicularis and Corrugator injections

SUMMARY:
The purpose of this study is to describe three safe and reproducible techniques for brow lifting using botulinum toxin. It will also describe the effect of 2 techniques on the eyebrow shape using quantitative, objective measurements and satisfaction scales.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive 30 female patients presenting to our clinic for brow lifting with botulinum toxin will be randomized to receive one of the two injection techniques

Exclusion Criteria:

* Patients with previous periorbital/forehead surgery
* Patients who plucked the upper eyebrow margin
* Patients with eyebrow tatoos
* Patients with upper face botulinum toxin injection in the past 12 months
* Patients with resorbable upper face fillers injection in the past 12 months
* Patients with previous permanent upper face fillers injection
* Pregnant patients
* Lactating patients
* Patients with preexisting neuromuscular conditions (myasthenia gravis, Eaton Lambert syndrome)
* Patients using medication that could potentiate the effect of botulinum (ex: aminoglycoside antibiotics)
* Patients with sensitivity to botulinum toxin or human albumin

Ages: 28 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Objective assessment | 15 days post treatment
  Objective assessment will be done on anteroposterior views of pre-and-post injection photographs. The mid pupillary line will be drawn and the eyebrow vertical height will be measured from this line to the upper border of the brow at seven horizontal points: the most medial aspect of the eyebrow, medial canthus, medial limbus, mid pupil, lateral limbus, lateral sclera, and most lateral eyebrow.

SECONDARY OUTCOMES:
Patient satisfaction | 15 days post treatment
  Patient satisfaction will be determined by a questionnaire completed at 15 days post-treatment. Subjects will indicate how satisfied they are on a 4-point scale (1-4) as follow:
  1. Very Satisfied
  2. Satisfied
  3. Dissatisfied
  4. Very Dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu De France, Beirut, Aschrafieh, Lebanon

REFERENCES:
- [Derived] El-Khoury JS, Jabbour SF, Awaida CJ, Rayess YA, Kechichian EG, Nasr MW. The Impact of Botulinum Toxin on Brow Height and Morphology: A Randomized Controlled Trial. Plast Reconstr Surg. 2018 Jan;141(1):75-78. doi: 10.1097/PRS.0000000000003919. PMID 29280866